CLINICAL TRIAL: NCT03249480
Title: Pegylated Somatropin (PEG Somatropin) in the Treatment of Children With Growth Hormone Deficiency: A Multicenter, Open-label, Phase IV Clinical Trial With Different Administration Dosage of PEG Somatropin
Brief Title: Pegylated Somatropin (PEG Somatropin) in the Treatment of Children With Growth Hormone Deficiency
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Collaborators: Beijing Children's Hospital (Other); Tianjin Medical University General Hospital (Other); Peking University Third Hospital (Other); China-Japan Friendship Hospital (Other); Dalian Children's Hospital (Other); Xian Children's Hospital (Other Government); Wuhan Children's Hospital (Other); Fuzhou Children s Hospital (Unknown); Anhui Provincial Children's Hospital (Other); Hunan Children's Hospital (Other Government); Shenzhen Children's Hospital (Other Government); Children's Hospital of Hebei Province (Other); Second Affiliated Hospital of Xi'an Jiaotong University (Other); Zhengzhou Children's Hospital, China (Other); Children's Hospital of Soochow University (Other); Maternal and Child Health Hospital of Guangxi Zhuang Autonomous Region (Other); First Affiliated Hospital of Kunming Medical University (Other); Kunming Children's Hospital (Other); The First People's Hospital of Yunnan (Other); Xuzhou Children's Hopspital (Unknown); Henan Provincial People's Hospital (Other); The First Affiliated Hospital of Henan University of Traditional Chinese Medicine (Other); First Affiliated Hospital of Harbin Medical University (Other); The Second Hospital of Hebei Medical University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Union Hospital of Tongji Medical College of HUST (Unknown); Wuxi Women's & Children's Hospital (Other); The Second Affiliated Hospital of Kunming Medical University (Other); Nanjing Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GenSci 004 CT-GCX
Record Dates: First submitted 2017-07-24; First posted 2017-08-15 (Actual); Last update posted 2017-08-15 (Actual); Status verified 2017-07

CONDITIONS: Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEG-somatropin (Experimental): 30IU/10 mg/3ml/kit, 0.1-0.2mg /kg/w, once per day for 26 weeks.
  Interventions: Biological: PEG-somatropin

INTERVENTIONS:
Biological: PEG-somatropin — 30IU/10 mg/3ml/kit, 0.1-0.2mg /kg/w, once per day for 26 weeks.

SUMMARY:
To Evaluate the safety and efficacy of PEG Somatropin in the treatment of children with growth hormone deficiency, as well as to study the dosage of PEG Somatropin.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as GHD before starting treatment, according to medical history, clinical symptoms and signs, GH provocation tests and imaging and other examinations:

  1. According to statistical height data of physical development of Chinese children in nine cities in 2005, the height is lower than 3rd percentile growth curve of the same age, same sex normal children;
  2. Height velocity (HV) ≤5.0 cm / yr;
  3. GH provocative tests (with two drugs of different mechanism of action) confirmed plasma GH peak <10.0 ng / ml;
  4. bone age for girl≤9 years old, for Boy≤10 years old, bone age is one year or more later than the actual age, that is the actual age - bone age ≥ 1 year;
* Before puberty (Tanner I stage), age≥3 years old, male or female;
* Have not received hormone therapy within 6 months;
* Subjects is willing and able to cooperate to complete scheduled visits, treatment plans and laboratory tests and other procedures, to sign informed consent.

Exclusion Criteria:

* Dysfunction of liver and kidney (ALT> 2 times the upper limit of normal, Cr> upper limit of normal);
* Patients positive for hepatitis B c-antibody (HBcAb), hepatitis B surface antigen (HBsAg) or hepatitis B e antigen (HBeAg);
* Patients with known hypersensitivity to PEG Somatropin or Somatropin or any other components of the study product;
* Patients with severe cardiopulmonary or hematological diseases, a current or past history of malignant tumors, immunodeficiency diseases, or mental diseases;
* Potential cancer patients (family history);
* Patients with diabetics;
* Patients with other growth disorders, such as Turner's syndrome, sexual physical delayed puberty, Laron syndrome, growth hormone receptor deficiency, girls with slowly growing who did not rule out chromosomal abnormalities;
* Patients with congenital bone dysplasia or scoliosis;
* Subjects took part in other clinical trial study during 3 months;
* Other conditions in which the investigator preclude enrollment into the study.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 900 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Ht SDSca (Height Standard Deviation Score for Chronological Age) | Baseline
  Ht SDSca was calculated by dividing the difference between the actual height of a patient and the mean height of the population for that chronological age by the standard deviation (SD) of the height of the population for that chronological age
Change of yearly growth velocity from baseline to 26 weeks | Baseline, 26 weeks after initiating treatment
  Height velocity calculate by formula
Ht SDSca | 26 weeks after initiating treatment
  Ht SDSca was calculated by dividing the difference between the actual height of a patient and the mean height of the population for that chronological age by the standard deviation (SD) of the height of the population for that chronological age

SECONDARY OUTCOMES:
Ht SDSBA (Height Standard Deviation Score for Bone Age) | Baseline,26 weeks after initiating treatment
IGF-1 SDS (IGF-1 Standard Deviation Score) | Baseline,26 weeks after initiating treatment
IGFBP-3 SDS (IGFBP-3 Standard Deviation Score) | Baseline,26 weeks after initiating treatment
Skeletal maturity | Baseline,26 weeks after initiating treatment
  Skeletal maturity=(Bone Age at 26 weeks-Bone Age at baseline)/treatment duration

CONTACTS AND LOCATIONS:
Overall Officials: Chunxiu Gong, Principal Investigator — Beijing Children's Hospital
Locations (28):
- China (28):
  - Anhui Provincial Children's Hospital, Hefei, Anhui
  - Fuzhou Children s Hospital, Fuzhou, Fujian
  - Sun Yat-Sen Memorial Hospital, Guangzhou, Guangdong
  - The Second Hospital of Hebei Medical University, Shijiangzhuang, Hebei
  - Children's Hospital of Hebei Province, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Children's Hospital of Zhengzhou, Zhengzhou, Henan
  - Henan Provincal People's Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Henan University of TCM, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, HUST, Wuhan, Hubei
  - Wuhan Children's Hospital, Wuhan, Hubei
  - Hunan Children's Hospital, Changsha, Hunan
  - Maternal & Child Health Hospital of Guangxi Zhuang Autonomous Region, Nanjing, Jiangsu
  - Nanjing Children's Hospital, Nanjing, Jiangsu
  - Children's Hospital of Soochow University, Suzhou, Jiangsu
  - Wuxi Children's Hospital, Wuxi, Jiangsu
  - Xuzhou Children's Hpspital, Xuzhou, Jiangsu
  - Dalian Children's Hospital, Dalian, Liaoning
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Xi'an Children's Hospital, Xi’an, Shanxi
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Kunming Children's Hospital, Kunming, Yunnan
  - Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The First People's Hospital of Yunnan Province, Kunming, Yunnan
  - China-Japan Friendship Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Shenzhen Children's Hospital, Shenzhen
  - Tianjin Medical University General Hospital, Tianjin

REFERENCES:
- [Derived] Chen J, Zhong Y, Wei H, Chen S, Su Z, Liu L, Liang L, Lu P, Chen L, Chen R, Ni S, Wang X, Li L, Wang Y, Xu X, Xiao Y, Yao H, Liu G, Jin R, Cao B, Wu D, Su C, Li W, Qin M, Li X, Luo X, Gong C. Polyethylene glycol recombinant human growth hormone in Chinese prepubertal slow-growing short children: doses reported in a multicenter real-world study. BMC Endocr Disord. 2022 Aug 9;22(1):201. doi: 10.1186/s12902-022-01101-8. PMID 35945517